CLINICAL TRIAL: NCT03041298
Title: Evaluation of Efficacy and Safety of Dotarem in Magnetic Resonance Mammography
Brief Title: Post Marketing Surveillance Study for Evaluation of Efficacy and Safety of Dotarem in Magnetic Resonance Mammography
Status: Completed | Type: Observational
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Other Study IDs: DGD-55-006
Record Dates: First submitted 2017-02-01; First posted 2017-02-02 (Estimated); Results first posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-03

CONDITIONS: MR Mammography With Dotarem
MeSH Terms: interventions — gadoterate meglumine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All included patients: All included patients underwent MR mammography with Dotarem
  Interventions: Procedure: MR mammography with Dotarem

INTERVENTIONS:
Procedure: MR mammography with Dotarem
  Other Names: MR mammography with gadoteric acid/gadoterate meglumine

SUMMARY:
Guerbet conducted a non-interventional post-marketing surveillance study on its Magnetic Resonance Imaging (MRI) contrast agent Dotarem (gadoteric acid/gadoterate meglumine) from September 2011 to December 2013. The aim of this study, which was conducted in accordance with section 67, paragraph 6 of the German drug regulation, Arzneimittelgesetz, was to generate additional data on the diagnostic efficacy, reliability and safety of Dotarem in Magnetic Resonance (MR) mammography.

DETAILED DESCRIPTION:
Diagnostic efficacy was assessed on the basis of image quality (5-stage scale from "excellent" to "very poor"), diagnosis and cytology test result. Safety was assessed on the basis of the frequency and seriousness of adverse drug reactions observed following the injection of Dotarem.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for high-resolution MR mammography using the MRI contrast agent Dotarem

Exclusion Criteria:

-

Max Age: 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric patients who are scheduled for high-resolution MR mammography using the MRI contrast agent Dotarem
Sampling Method: Non-Probability Sample
Enrollment: 1537 (Actual)
Dates: Start 2011-09; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Included Patients
Started | 1537
Completed | 1537
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Included Patients
Number analyzed (Participants) | 1537
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (12.3)
Age, Customized [Count of Participants; unit: Participants]
  <25 years | 8
  between 25 and 55 years | 1025
  >55 years | 504
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender was missing for 43 patients.
  Participants
    number analyzed (Participants) | 1494
    Female | 1491
    Male | 3
Menopausal status [Count of Participants; unit: Participants] — Menopausal status was recorded before MR mammography. Population: Menopausal status was missing for 31 patients.
  Participants
    Premenopausal: number analyzed (Participants) | 1506
    Premenopausal | 506
    Perimenopausal: number analyzed (Participants) | 1506
    Perimenopausal | 174
    Postmenopausal: number analyzed (Participants) | 1506
    Postmenopausal | 826
Risk factors [Count of Participants; unit: Participants] — Risk factors were recorded before MR mammography. Population: Risk factors were missing for 270 patients.
  Participants
    Family history: number analyzed (Participants) | 1267
    Family history | 428
    Personal history: number analyzed (Participants) | 1267
    Personal history | 525
    Family and personal history: number analyzed (Participants) | 1267
    Family and personal history | 300
    Other: number analyzed (Participants) | 1267
    Other | 14

OUTCOME MEASURES:

1. Primary Outcome: Image Quality
Description: Image quality was evaluated on a 5-point scale: "excellent"; "good"; "moderate"; "poor" and "very poor".
Time Frame: During MRI procedure
Population: Image quality was missing for 16 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | All Included Patients
Number analyzed (Participants) | 1521
Participants
  Excellent | 495
  Good | 898
  Moderate | 118
  Poor | 8
  Very Poor | 2

2. Primary Outcome: Ability to Make a Diagnosis
Description: Ability to make a diagnosis was evaluated by answering "yes" or "no" to the question "Did the examination permit a diagnosis ?"
Time Frame: During MRI procedure
Population: Ability to make a diagnosis was missing for 2 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | All Included Patients
Number analyzed (Participants) | 1535
Participants
  Yes | 1523
  No | 12

3. Primary Outcome: Diagnostic Results (Percentage of Patients Per Diagnosis)
Description: Diagnoses were made with MR images. Percentage of patients per diagnosis was calculated. Multiple diagnoses were possible for the same patient.
Time Frame: During MRI procedure
Population: Diagnosis was achieved in 1523 patients but results were missing for 4 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | All Included Patients
Number analyzed (Participants) | 1519
Participants
  Benign changes | 858
  Normal findings | 324
  Unilateral focal pathological findings | 159
  Other | 101
  Invasive ductal carcinoma | 72
  Bilateral focal pathological findings | 23
  Carcinoma in situ | 12
  Extensive intraductal component | 7

4. Primary Outcome: Cytology Test Results (Percentage of Patients Per Cytology Test Result)
Description: Diagnoses were made according to the cytology test results. Percentage of patients per cytology test result was calculated. Multiple diagnoses were possible for the same patient.
Time Frame: During MRI procedure
Population: A cytology test was performed in 232 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | All Included Patients
Number analyzed (Participants) | 232
Participants
  Invasive ductal carcinoma | 109
  Other | 66
  Invasive lobular carcinoma | 35
  Intraductal carcinoma | 14
  Fibroadenoma | 8
  Mucinous carcinoma | 3
  Inflammatory carcinoma | 2
  Papilloma | 2
  Medullary carcinoma | 1
  Invasive papillary carcinoma | 1
  Tubular carcinoma | 1

5. Primary Outcome: Frequency of Adverse Drug Reactions
Description: The frequency of adverse drug reactions (serious and non-serious) that occurred following injection of Dotarem was recorded. Adverse drug reactions are adverse events related to the product administered.
Time Frame: From the beginning of the MR mammography procedure to 30-60 min after
Measure: Number; unit: Adverse drug reactions
Arm/Group | All Included Patients
Number analyzed (Participants) | 1537
Adverse drug reactions | 12

ADVERSE EVENTS:
Time Frame: From the beginning of the MR mammography procedure to 30-60 min after
Description: Adverse events reported were related to the product administered. Several adverse events could be reported for the same patient.
Arm/Group | All Included Patients
All-Cause Mortality (participants affected / at risk) | 0/1537
Serious Adverse Events (participants affected / at risk) | 1/1537
Other Adverse Events (participants affected / at risk) | 4/1537
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Included Patients (N=1537)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Included Patients (N=1537)
Palpitations (Cardiac disorders) | 1 (1)
Vomiting projectile (Gastrointestinal disorders) | 1 (1)
Feeling hot (General disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No